CLINICAL TRIAL: NCT05297656
Title: The Effect of Instrument Assisted Soft Tissue Mobilization in Female Patients With Myofascial Pain Syndrome Due to Active Trigger Points in the Upper Trapezius Muscles
Brief Title: The Effect of Instrument Assisted Soft Tissue Mobilization in Female Patients With Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, Assistant professor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-77504701-604.02.-00000386201; Local ethics (Other: 2022-03/21)
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Myofascial Pain; Instrument Assisted Soft Tissue Mobilization
Keywords: miyofascial pain; Instrument Assisted Soft Tissue Mobilization; Quality of life

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: This study was designed as blinded, randomized and controlled. The person who evaluates the patients before and after the treatment is blind. In other words, the person evaluating the patients and the person giving the treatment are different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Group (Experimental): A total of 8 sessions of graston massage protocol will be applied to the patients in the experimental group for 4 weeks, 2 days a week for 5 minutes, at the hospital operating within the body of Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center.
  All patients will also receive home exercise therapy including stretching of the trapezius muscle and posture exercises
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization; Other: Home exercises programe
- Sham Comparator Group (Sham Comparator): A total of 8 sessions of sham graston massage protocol will be applied to the patients in the experimental group for 4 weeks, 2 days a week for 5 minutes, at the hospital operating within the body of Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center.
  Sham graston massage is not a deep tissue massage, but will be performed with the device superficially, without applying pressure and mobilization.
  All patients will also receive home exercises.
  Interventions: Other: Sham Instrument Assisted Soft Tissue Mobilization; Other: Home exercises programe
- Control group (Other): The volunteers in the control group will be only given home exercise therapy including stretching of the trapezius muscle and posture exercises
  Interventions: Other: Home exercises programe

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — Instrument Assisted Soft Tissue Mobilization with graston tecnique and Home exercises programe
  Arms: Experimental Group
Other: Sham Instrument Assisted Soft Tissue Mobilization — Instrument Assisted Soft Tissue Mobilization to be applied superficially so it is not like a real graston tecnique and Home exercises programe
  Arms: Sham Comparator Group
Other: Home exercises programe — Only Home exercises programe

SUMMARY:
The primer aim of this study is to demonstrate the effecti of instrument assisted soft tissue mobilization on pain, functionality, quality of life and depression in the treatment of female patients with myofascial pain syndrome due to active trigger points in the upper trapezius muscles

DETAILED DESCRIPTION:
Myofascial Pain Syndrome (MAS); It is a non-articular, non-inflammatory regional musculoskeletal pain syndrome characterized by myofascial trigger points located at muscle, fascia or tendon insertion sites and the spread of pain to reference areas by palpation of these points.

h The effectiveness of massage therapy in MAS is known. In this study, investigators will apply instrument assisted deep tissue mobilization (graston massage). Instrument-assisted soft tissue mobilization massage, which is a type of massage, will be applied by a physiotherapist who has a certificate on this subject and takes part as an assistant researcher in our study.

Soft tissue mobilization is a unique soft tissue mobilization combined with active mobility and stretching exercises already prescribed for patients with musculoskeletal injuries.

The various sizes and beveled edges of the stainless steel instruments allow physiotherapists to tailor treatment to different muscle structures facing myofascial constraints.

Localized increases in blood flow and soft tissue realignment lead to muscle function, increased normal joint motion, and decreased pain.

It has been investigated in the literature for many different diseases (trigger finger, nonspecific low back pain, myofascial pain syndrome) and found to be effective.CF

ELIGIBILITY:
Inclusion Criteria:

1. Being woman and between the ages of 18-45
2. Not to be in menopause
3. Pain in the upper trapezius area
4. Detection of a taut band in the upper trapezius region on examination
5. At least one active trigger point in the tension band in the upper trapezius region on examination
6. The pain caused by the compression of the trigger point is the pain that the patient complains about
7. Painful restriction of cervical lateral flexion motion during stretching
8. Pain 4 or more according to NRS

Exclusion Criteria:

1. major surgery or trauma to the musculoskeletal system, especially the spine and upper extremities 2.History of any operation related to the head and neck region 3. Neuromuscular disease 4. History of rheumatic disease, malgnite in the active period 4. Cervical discopathy, cervical spondylosis, pathologies related to the shoulder joint and surrounding soft tissues, scoliosis, kyphosis, leg length difference, polio sequelae, developmental hip dysplasia 5. Psychiatric disease (Beck Depression Inventory score of 30 and above) 6.Obese (BMI≥30 kg/m2)

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since the anatomical muscle structure and physiology of men and women are different, we only made it in women in order to eliminate this difference.
Enrollment: 75 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Pain Algometer | Baseline
  The pain threshold level will be measured with an algometer. The algometer manually evaluates the patient's pain threshold and gives a numerical data
Pain Algometer | Fourth week (Posttreatment)
  The pain threshold level will be measured with an algometer. The algometer manually evaluates the patient's pain threshold and gives a numerical data
Visual Analogue Scale (VAS) | Baseline
  Visual Analogue Scale (VAS) for pain assessment. In this scale, which evaluates pain with a 10-point Likert scale, 0 is scored as no pain, 5 as moderate pain, and 10 as excruciating pain.
Visual Analogue Scale (VAS) | Fourth week (Posttreatment)
  Visual Analogue Scale (VAS) for pain assessment. In this scale, which evaluates pain with a 10-point Likert scale, 0 is scored as no pain, 5 as moderate pain, and 10 as excruciating pain.
Number and location of trigger points | Baseline
  The number and location of trigger points that cause myofascial pain will be determined and recorded by examination.
Number and location of trigger points | Fourth week (Posttreatment)
  The number and location of trigger points that cause myofascial pain will be determined and recorded by examination.

SECONDARY OUTCOMES:
Beck depression questionnaire | Baseline
  Beck depression questionnaire is a questionnaire consisting of 21 questions that evaluates the mood of the patient and has Turkish validity and reliability(1).
Beck depression questionnaire | Fourth week (Posttreatment)
  Beck depression questionnaire is a questionnaire consisting of 21 questions that evaluates the mood of the patient and has Turkish validity and reliability(1).
The World Health Organization health-related quality of life-brief form | Baseline
  The World Health Organization health-related quality of life-brief form (WHO-health-related quality of life-brief form)
The World Health Organization health-related quality of life-brief form | Fourth week (Posttreatment)
  The World Health Organization health-related quality of life-brief form (WHO-health-related quality of life-brief form)
The neck disability index | Baseline
  The neck disability index is a questionnaire consisting of 10 questions with Turkish validity and reliability, which recognizes the functional evaluation of neck pain (3). Each question is scored between 0 and 5. High scores are associated with increased disability.
The neck disability index | Fourth week (Posttreatment)
  The neck disability index is a questionnaire consisting of 10 questions with Turkish validity and reliability, which recognizes the functional evaluation of neck pain (3). Each question is scored between 0 and 5. High scores are associated with increased disability.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Asst Prof, Study Director — university
Locations (1):
- Kırşehir Ahi Evran University Faculty of Medicine, Kırşehir, City Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No